CLINICAL TRIAL: NCT06149949
Title: Ambispective Pilot Study on the Prevalence of Chronic Rhinosinusitis Associated With Inflammatory Bowel Disease and Association With Biomarkers of Epithelial Barrier Damage
Brief Title: the Prevalence of Chronic Rhinosinusitis Associated With Inflammatory Bowel Disease and Association With Biomarkers of Epithelial Barrier Damage
Acronym: PRIME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6126
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Intestinal Inflammation; Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — the aim of the study is to define the prevalence of rhinosinusitis cronic in intestinal bowel disease patients, to assess how it affects the patient's quality of life, and any correlations between these two entities

SUMMARY:
The goal of this observational study is to define the prevalence of chronic rhinosinusitis in patients with intestinal bowel disease.

The main questions it aims to answer are:

* Evaluate the influence of chronic rhinosinusitis on the quality of life of patients with intestinal bowel disease
* Evaluate any relationships between chronic rhinosinusitis and the clinical course of intestinal bowel disease -Evaluate the influence of chronic rhinosinusitis on the response to biologic therapies for intestinal bowel disease
* Evaluate mucosal barrier damage in patients with chronic rhinosinusitis and intestinal bowel disease by collecting blood and stool samples according to clinical practice
* Presence of enterotoxin sensitization to S. Aureus in patients with intestinal bowel disease
* Histopathological evaluation: reevaluation of biopsy slides performed according to clinical practice will be performed in patients with chronic rhinosinusitis and intestinal bowel disease in order to quantify the proportion of eosinophilic infiltrate at the intestinal level and to assess any differences from the population with intestinal bowel disease only.

Patients with intestinal bowel disease afferent to our outpatient chronic inflammatory bowel disease clinic at CEMAD will be enrolled.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Age between 18 years and 70 years.
* Diagnosis of Crohn's disease or Ulcerative Rectocolitis
* Willingness to participate in the study and ability to comply with and understand the study protocol.
* Patients with a previous diagnosis of Crohn's disease or Ulcerative Rectocolitis for at least 3 months prior to screening
* Signature of informed consent

Exclusion Criteria:

* Age <18 years
* Refusal of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intestinal bowel disease afferent to our outpatient chronic inflammatory bowel disease clinic at CEMAD will be enrolled. All patients will be given questionnaires at baseline on quality of life and symptoms of intestinal bowel disease and the presence of symptoms correlated with rhinosinusitis cronic. Patients who respond affirmatively to the presence of rhinosinus symptoms will have their blood drawn according to clinical practice and deliver a stool sample for gut microbiota analysis. In addition, all will undergo psychological evaluation. Patients with rhinosinusitis cronic will undergo specialist otolaryngologist evaluation according to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of chronic rhinosinusitis in patients with chronic inflammatory bowel disease | 1 hour
  To define the prevalence of chronic rhinosinusitis in patients with chronic inflammatory bowel disease